CLINICAL TRIAL: NCT05277909
Title: Effectiveness of an Expert Assessment and Individualised Treatment in Comparison to a Minimal Home-based Exercise Program in Women With Late-term Shoulder Impairments After Primary Breast Cancer Surgery.
Brief Title: An Individualised Treatment vs. a Minimal Program in Women With Late-term Shoulder Impairments After Breast Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Region of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-20200021, 19-16321
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Shoulder Pain; Late Effect; Breast Cancer; Rehabilitation
Keywords: Shoulder Impairments; Late Term; Breast Cancer; Rehabilitation
MeSH Terms: conditions — Shoulder Pain; Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The expert assessment of shoulder impairments and individualised treatment plan (Experimental): Participants randomised to the Intervention group will be referred to an expert assessment of their shoulder impairments at the Shoulder Sector, Vejle Hospital - Orthopaedic Department. The expert assessment will be performed by experienced specialists (e.g. physician and physiotherapist) who are specialised in shoulder diagnostics using x-ray, ultrasound, anamnesis/history and standard clinical tests such as Neers, Hawkins, Jobe´s Empty Can, Painful Arc and Resisted External Rotation. The participant's diagnosis based on the history, symptoms and clinical findings will be used to guide the individualised treatment plan. The individualised treatment plan will typically contain a referral to physiotherapeutic treatment at the municipality or private practice, receive specialised physiotherapeutic rehabilitation at Vejle Hospital, get an ultrasound guided corticosteroid injection in the shoulder or offer surgery.
  Interventions: Other: The expert assessment of shoulder impairments and individualised treatment plan
- A minimal physiotherapeutic rehabilitation program delivered in a pamphlet (Active Comparator): Participants randomised to the Control comparator group will receive a pamphlet from the secretary and perform the exercises at home. This pamphlet contains a program with minimal exercise recommendations for the shoulder consisting of mobility, stretching, strength exercises and tissue treatment. The purpose is to stimulate circulation, improve shoulder function (mobility), increase muscle strength and reduce shoulder pain. The program consists of three warm-up exercises (arm swing, shoulder rolling and scapula-back pocket exercise) followed by three stretching exercises for the breast and shoulder area. Furthermore the pamphlet includes a tissue treatment and four strength exercises for the shoulder (external rotation, extension and flexion of the shoulder and diagonal pull apart). Mobility (with 5-10 repetitions), stretching exercises (in 30 seconds) and tissue treatments will be performed twice a day, while the strength exercises will be performed once a day with 3x12 repetitions.
  Interventions: Other: A minimal physiotherapeutic rehabilitation program delivered in a pamphlet

INTERVENTIONS:
Other: The expert assessment of shoulder impairments and individualised treatment plan — The participant's diagnosis based on the history, symptoms and clinical findings will be used to guide the individualised treatment plan.
  Arms: The expert assessment of shoulder impairments and individualised treatment plan
Other: A minimal physiotherapeutic rehabilitation program delivered in a pamphlet — This pamphlet contains a program with minimal exercise recommendations for the shoulder consisting of mobility, stretching, strength exercises and tissue treatment.
  Arms: A minimal physiotherapeutic rehabilitation program delivered in a pamphlet

SUMMARY:
In breast cancer patients late-term upper limb sequelae, such as shoulder pain and impaired shoulder function remain common after primary breast cancer surgery. The aim of this trial is to evaluate whether an expert assessment of shoulder impairments, followed by an individualised treatment plan, is superior to a minimal physiotherapeutic rehabilitation program in reducing shoulder symptoms, assessed 12 weeks after initiation of treatment, among women with late-term shoulder impairments after primary breast cancer surgery.

DETAILED DESCRIPTION:
Worldwide, breast cancer is the second most common cancer. Internationally, an age-standardised incidence rate between 83.1 and 111.9 per 100.000 women is seen, with Denmark taking an unfortunate second place. Standard surgical treatment in Denmark is breast-conserving surgery (BCS) or mastectomy in combination with sentinel lymph node dissection (SLND) or axillary lymph node dissection (ALND). In part due to early diagnosis and optimised treatment methods, 5-year survival has improved to a current 87%. Despite fewer mastectomies and more BCS, less invasive surgical procedures of the axilla (e.g. fewer ALND vs. SLND), and more refined radiotherapy procedures, late-term upper limb impairment still remains common. The most frequent are lymphoedema, sensory disturbances, pain and impaired shoulder function, with up to 70% of patients reporting at least one of these symptoms three years after surgery. These impairments lead to difficulties in activities of daily living, increased risk of depression and anxiety and decreased quality of life (QoL).

Previous research has primarily focused on prevention and treatment of lymphedema, and less on other upper limb impairments. Pre- and early postoperative physiotherapeutic interventions are known to be effective in reducing shoulder pain and improving shoulder function after breast cancer treatment. Nonetheless, late-term upper limb impairments need further focus with prevalence´s of up to 50% is reported for impaired shoulder function and pain up to 6 years after surgery, and a substantial knowledge gap exists as to how to help these women. Currently, no standardised evaluation of their impairments or treatment is offered, and it is therefore up to the individual woman to seek care, resulting in large variations in rehabilitation. Thus a substantial knowledge gap exists in how to meet the rehabilitation needs of these women and evaluation of the actual burden of late-term shoulder impairments after primary treatment for breast cancer and the effect of different treatment strategies is warranted.

The primary aim of this study is to investigate whether the effect of a patient-centred specialised intervention, consisting of an expert assessment followed by an individualised treatment plan (i.e. Intervention group), is superior to a minimal physiotherapeutic rehabilitation program delivered in a pamphlet (i.e. Control comparator group) among women with late-term shoulder impairments 3-7 years after their primary breast cancer surgery. The hypothesis is that women randomised to the Intervention Group will improve significantly more in shoulder function and pain 12 weeks after initiating the treatment than those randomised to the Control comparator group.

This trial is a stratified (by type of surgery and radiotherapy), block randomised (1:1 allocation), controlled, parallel group and assessor blinded superiority trial conducted in Denmark. 130 participants with late-term shoulder impairments 3-7 years after primary surgery for breast cancer will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer patients who underwent unilateral BCS or mastectomy on the left or right side, including SLND or +/- ALND within the last 3-7 years (2015-2019)
2. Currently living in the Region of Southern Denmark or Central Denmark Region with a radius of 75 km from Vejle Hospital
3. Between 18 and 71 age on time of surgery for primary breast cancer
4. Indicate pain in chest and/or shoulder area (shoulder impairments) as the biggest problem/late-term effect in everyday life
5. Indicate impaired shoulder function due to pain or due to tightness/tension
6. Indicate shoulder pain at rest, during general activities, during sleep or during flexion, rotation or abduction of the shoulder
7. A score ≥15 on the Disabilities of the Arm, Shoulder and Hand (Quick DASH)
8. Agree to participate in this trial and signs written informed consent

Exclusion Criteria:

1. No previous breast cancer (before 2014)
2. Cancer relapse after the date of index surgery, cancer spread outside of thorax and axilla, tumor fixed to chest wall
3. Primary- or secondary breast reconstruction performed at any time
4. Severe lymphedema (an average score ≥ 70% in the first 7 questionnaires on the LYMPH-ICF-DK
5. Bilateral breast cancer surgery
6. Previous surgery in the affected shoulder (prior to inclusion)
7. Previous shoulder or upper limb fractures (left/right)
8. Currently receiving chemo, immuno- or radiotherapy
9. Co-morbidity expected to influence shoulder function (e.g. rheumatoid arthritis, previous stroke, multiple sclerosis)
10. Other reasons for exclusion (e.g. pregnancy, not legally competent, unable to comprehend the information or unable to consent)

Ages: 18 Years to 78 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Change in Shoulder Pain and Disability Index (SPADI) from baseline to 12 weeks after initiating the treatment. | 0, 4, 8 and 12 weeks
  SPADI is a 13-item patient-reported outcome measure to assess shoulder pain (5 items) and shoulder function (8 items) within the last week. The items are scored on a numeric rating scale that ranges from 0 (no pain/no difficulty) to 10 (worst pain/so difficult that required help). Each domain score is equally weighted and added to a total percentage score that ranges from 0 (best) to 100 (worst). The higher the score, patients reported shoulder impairments. The region specific questionnaire can be used in patients with different or unspecified shoulder diagnoses. SPADI is valid, reliable and responsible measure among patients with shoulder impairments.

SECONDARY OUTCOMES:
Change in SPADI pain from baseline to 12 weeks after initiating the treatment. | 0, 4, 8 and 12 weeks
  Change in SPADI pain will be reported as a separate subscale. The 5-item pain subscale are scored on a numeric rating scale that ranges from 0 (no pain) to 10 (worst pain). The higher the score, patients report greater shoulder pain and reduction in the SPADI pain score will suggest improvement.
Change in SPADI function from baseline to 12 weeks after initiating the treatment. | 0, 4, 8 and 12 weeks
  Change in SPADI function will be reported as a separate subscale. A 6-item version (exclusion of question three and seven) of the disability subscale exhibited adequate fit in the Danish version. The 6-item disability subscale are scored on a numeric rating scale that ranges from 0 (no difficulty) to 10 (so difficult that required help). The higher the score, patients report greater shoulder disabilities and reduction in the SPADI function score will suggest improvement.
SPADI clinical response. | 12 weeks (follow-up)
  Response to treatment will be computed for the SPADI change score for each woman in both treatment groups and presented dichotomised (i.e. responder and non-responder) as number (and percentages) responders. Women will be classified as an responder if the SPADI change score improves by 8 points or more (≥), corresponding to the minimal clinically important difference on SPADI from baseline to 12 weeks follow-up.
Global Perceived Effect (GPE) measured at 4, 8 and 12 weeks after initiating the treatment. | 4, 8 and 12 weeks
  The GPE will evaluate the impression of the treatment's success including overall shoulder problems on a 7-point Likert scale ranging from "markedly worse" to "markedly improved".
Change in Active Range Of Motion (A-ROM) in the affected shoulder from baseline to 12 weeks after initiating the treatment. | 0 and 12 weeks
  A smartphone inclinometer (GetMyROM) will be used to assess A-ROM in flexion, internal rotation, external rotation and abduction respectively the operated side. After one test trial, the mean value of three measurements will be taken for both flexion, rotation and abduction respectively the operated side.
Change in Passive Range Of Motion (P-ROM) in the affected shoulder from baseline to 12 weeks after initiating the treatment. | 0 and 12 weeks
  A smartphone inclinometer (GetMyROM) will be used to assess P-ROM in flexion, internal rotation, external rotation and abduction respectively the operated side. After one test trial, the mean value of three measurements will be taken for both flexion, rotation and abduction respectively the operated side.
Number of treatments received due to shoulder symptoms from baseline to 12 weeks after initiating the treatment. | 12 weeks (follow up)
  Number of visits to a healthcare professional (e.g. physician, chiropractor or physiotherapist) at hospital, municipality rehabilitation or private practice due to the shoulder symptoms during the intervention period, will be collected by using a patient-reported questionnaire.
Change in maximum shoulder pain intensity within the previous 24 hours in the affected shoulder measured by Numeric Rating Scale (NRS) from baseline to 12 weeks after initiating the treatment. | 0, 4, 8 and 12 weeks
  The NRS pain scale is a single 11-item patient reported outcome measure used to assess the maximum shoulder pain intensity. The scale ranges from 0 (no pain) to 10 (worst pain imaginable). The higher the score, patients report greater shoulder pain intensity and reduction in the NRS score will suggest improvement. The NRS is a reliable, valid and responsive measure of pain in patients with cancer.
Change in shoulder pain during general activities within the previous 24 hours in the affected shoulder measured by Numeric Rating Scale (NRS) from baseline to 12 weeks after initiating the treatment. | 0, 4, 8 and 12 weeks
  The NRS pain scale is a single 11-item patient reported outcome measure used to assess pain during general activities. The scale ranges from 0 (no pain) to 10 (worst pain imaginable). The higher the score, patients report greater shoulder pain and reduction in the NRS score will suggest improvement. The NRS is a reliable, valid and responsive measure of pain in patients with cancer.
Change in shoulder pain at rest within the previous 24 hours in the affected shoulder measured by Numeric Rating Scale (NRS) from baseline to 12 weeks after initiating the treatment. | 0, 4, 8 and 12 weeks
  The NRS pain scale is a single 11-item patient reported outcome measure used to assess pain at rest. The scale ranges from 0 (no pain) to 10 (worst pain imaginable). The higher the score, patients report greater shoulder pain and reduction in the NRS score will suggest improvement. The NRS is a reliable, valid and responsive measure of pain in patients with cancer.
Change in shoulder pain during sleep within the previous 24 hours in the affected shoulder measured by Numeric Rating Scale (NRS) from baseline to 12 weeks after initiating the treatment. | 0, 4, 8 and 12 weeks
  The NRS pain scale is a single 11-item patient reported outcome measure used to assess pain during sleep. The scale ranges from 0 (no pain) to 10 (worst pain imaginable). The higher the score, patients report greater shoulder pain and reduction in the NRS score will suggest improvement. The NRS is a reliable, valid and responsive measure of pain in patients with cancer.
Change in shoulder pain assessment during flexion/rotation/abduction in the affected shoulder measured by Numeric Rating Scale (NRS) from baseline to 12 weeks after initiating the treatment. | 0 and 12 weeks
  The NRS pain scale is a single 11-item patient reported outcome measure used to assess pain during flexion/rotation/abduction. The scale ranges from 0 (no pain) to 10 (worst pain imaginable). The higher the score, patients report greater shoulder pain and reduction in the NRS score will suggest improvement. The NRS is a reliable, valid and responsive measure of pain in patients with cancer.

OTHER OUTCOMES:
Change in pain medication consumption from baseline to 12 weeks after initiating the treatment. | 0, 4, 8 and 12 weeks
  Pain medication consumption in the past week due to shoulder related pain including questions about yes/no, type (prescription or nonprescription medicine) and frequency will be collected by using a patient-reported questionnaire.
Change in Patient Health Questionnaire - 9 (PHQ-9) from baseline to 12 weeks after initiating the treatment. | 0, 4, 8 and 12 weeks
  PHQ-9 is a 9-item patient-reported outcome measure to assess depression within the last 2 weeks. The total score ranges from 0 to 27; 5-9 = minimal symptoms, 10-14 = minor/mild depression, 15-19 = major depression, moderately severe, >20 = major depression, severe. The higher the score, patients report severe depression and reduction in the PHQ-9 score will suggest improvement. PHQ-9 is a reliable and valid measure of depression in cancer patients and the general population and can measure changes over time.
Change in General Anxiety Disorder - 7 (GAD-7) from baseline to 12 weeks after initiating the treatment. | 0, 4, 8 and 12 weeks
  GAD-7 is a 7-item patient-reported outcome measure to assess anxiety within the last 2 weeks. The total score ranges from 0 to 21; 0-4 = minimal anxiety symptoms, 5-9 = mild anxiety symptoms, 10-14 = moderate anxiety symptoms, >15 severe levels of anxiety symptoms. The higher the score, patients report severe anxiety and reduction in the GAD-7 score will suggest improvement. GAD-7 is a reliable and valid measure of anxiety in cancer patients and the general population.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Gordon Ingwersen, PT, PhD, Principal Investigator — Vejle Hospital
Locations (1):
- Department of Physio- and Occupational Therapy, Vejle Hospital, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Personal data for the primary and all secondary outcome measures will only be made available if required by the scientific journal, in which the result of the trial are published.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available after publication of the trial.
Access Criteria: Data access will be reviewed by the author group. Requestors will be required to sign a Data Access Agreement
URL: https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-022-06659-1

REFERENCES:
- [Derived] Feder KM, Lautrup MD, Nielsen SM, Egebaek HK, Rahr HB, Christensen R, Ingwersen KG. Effectiveness of an individualised treatment plan compared with a standard exercise programme in women with late-term shoulder impairments after primary breast cancer treatment: a randomised controlled trial. Acta Oncol. 2025 Mar 19;64:448-457. doi: 10.2340/1651-226X.2025.42737. PMID 40105684
- [Derived] Feder KM, Rahr HB, Lautrup MD, Egebaek HK, Christensen R, Ingwersen KG. Effectiveness of an expert assessment and individualised treatment compared with a minimal home-based exercise program in women with late-term shoulder impairments after primary breast cancer surgery: study protocol for a randomised controlled trial. Trials. 2022 Aug 20;23(1):701. doi: 10.1186/s13063-022-06659-1. PMID 35987857

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT05277909/SAP_000.pdf